CLINICAL TRIAL: NCT00289237
Title: A Randomised Non-pharmacological Intervention Study for Prevention of Ischaemic Heart Disease Inter99
Brief Title: Lifestyle Intervention in a General Population for Prevention of Ischaemic Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Birgitte Pickering, B. Pickering is the secretary of Professor Torben Joergensen, who is the primary investigator, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RCPH - 99-1
Record Dates: First submitted 2005-09-19; First posted 2006-02-09 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: CHD; AMI; CVD; Type 2 Diabetes; COLD
Keywords: Lifestyle intervention; Behavioural changes; CHD; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (3):
- High intensity intervention group (Experimental): Lifestyle intervention consisted of 15-30 minutes of individual lifestyle counselling + offer of participation in group-based lifestyle counselling (½ year). This offer was given at baseline to all participants in the group.
  Persons at high risk of IHD: offer additionally given at 1- and 3-year follow-up
  Interventions: Behavioral: Lifestyle intervention
- Low intensity intervention group (Experimental): Lifestyle intervention consisted of 15-30 minutes of individual lifestyle counselling. This offer was given at baseline to all participants in the group.
  Persons at high risk of IHD: offer additionally given at 1- and 3-year follow-up
  Interventions: Behavioral: Lifestyle intervention
- Control group (No Intervention): Questionnaires regarding lifestyle and general health were sent to all participants in this group.
  The importance of healthy lifestyle was not mentioned, and no intervention was offered.

INTERVENTIONS:
Behavioral: Lifestyle intervention
  Arms: High intensity intervention group; Low intensity intervention group

SUMMARY:
In spite of declining trend coronary heart disease (CHD) is still a leading cause of morbidity and mortality. Many years of epidemiological research have identified several risk factors for CHD. The main causes are physical inactivity and inappropriate diet (mediated through high blood pressure, high cholesterol and fatness) and smoking. So far intervention studies on lifestyle factors have shown disappointing results, most probably due to insufficient interventions and methodology.

Inter99 is a randomized non-pharmacological intervention study comprising 61,301 persons representing a well-defined population. About 13,000 are invited for a health examination and assessment of risk for CHD. Those at high risk are offered lifestyle intervention in three waves over a five year period. A priori the group is divided into a high intensive and low intensive intervention group. The remaining 48.285 individuals serve as control.

After five years all individuals who attended the base-line examination are re-invited to assess the effect of the intervention on intermediate end-points as lifestyle, absolute risk of CHD and biological risk factors. The total cohort (61.301) is followed through central registers to evaluate the effect of the intervention on use of the health care system and the long term effect on incidence of CHD.

The status for the project is that the four waves of intervention have been performed, the last follow-up was in March 2006.

Data collection finalized with 10 years follow-up via Central National Registries and a questionnaire. No further follow-up is scheduled for the main purposes of the study.

Analyses as regard the primary effect (on incidence of cardiovascular diseases) and secondary effect (on incidence of type 2 diabetes) are on-going. Analyses for a large number of spin off project are on-going.

More than 25 Ph.d. studies and more than 200 peer-review publication have so far been produced.

Summary of results, links to articles and theses at: www.Inter99.dk

DETAILED DESCRIPTION:
In spite of declining trend coronary heart disease (CHD) is still a leading cause of morbidity and mortality. Many years of epidemiological research have identified several risk factors for CHD. The main causes are physical inactivity and inappropriate diet (mediated through high blood pressure, high cholesterol and fatness) and smoking. So far intervention studies on lifestyle factors have shown disappointing results.

Inter99 is a randomized non-pharmacological intervention study comprising 61,301 persons representing a well-defined population. About 13,000 are invited for a health examination and assessment of risk for CHD. Those at high risk are offered lifestyle intervention in three waves over a five year period. A priori the group is divided into a high intensive and low intensive intervention group. The remaining 48.285 individuals serve as control.

After five years all individuals who attended the base-line examination are re-invited to assess the effect of the intervention on intermediate end-points as lifestyle, absolute risk of CHD and biological risk factors. The total cohort (61.301) is followed through central registers to evaluate the effect of the intervention on use of the health care system and the long term effect on incidence of CHD.

ELIGIBILITY:
Inclusion Criteria:

* All citizens in a predefined area

Exclusion Criteria:

* Drug abuse
* Language problem

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61301 (Actual)
Dates: Start 1999-03; Primary Completion 2006-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Incidence of CHD and other lifestyle related diseases after ten years | 2012
  Ongoing analyses in National Central Registers (Oct 2012)

SECONDARY OUTCOMES:
Changes in lifestyle and biological markers after one, three and five years | 2006
  Analyses completed. Results at: www.Inter99.dk

CONTACTS AND LOCATIONS:
Overall Officials: Torben Jørgensen, DrMedSci, Principal Investigator — Research Centre for Prevention and Health
Locations (1):
- Research Centre for Prevention and Health, Glostrup Municipality, Denmark

REFERENCES:
- [Background] Glumer C, Jorgensen T, Borch-Johnsen K; Inter99 study. Prevalences of diabetes and impaired glucose regulation in a Danish population: the Inter99 study. Diabetes Care. 2003 Aug;26(8):2335-40. doi: 10.2337/diacare.26.8.2335. PMID 12882858
- [Background] Husemoen LL, Thomsen TF, Fenger M, Jorgensen HL, Jorgensen T. Contribution of thermolabile methylenetetrahydrofolate reductase variant to total plasma homocysteine levels in healthy men and women. Inter99 (2). Genet Epidemiol. 2003 May;24(4):322-30. doi: 10.1002/gepi.10239. PMID 12687650
- [Background] Jorgensen ME, Glumer C, Bjerregaard P, Gyntelberg F, Jorgensen T, Borch-Johnsen K; Grennland Population Study. Obesity and central fat pattern among Greenland Inuit and a general population of Denmark (Inter99): relationship to metabolic risk factors. Int J Obes Relat Metab Disord. 2003 Dec;27(12):1507-15. doi: 10.1038/sj.ijo.0802434. PMID 14634682
- [Background] Jorgensen T, Borch-Johnsen K, Thomsen TF, Ibsen H, Glumer C, Pisinger C. A randomized non-pharmacological intervention study for prevention of ischaemic heart disease: baseline results Inter99. Eur J Cardiovasc Prev Rehabil. 2003 Oct;10(5):377-86. doi: 10.1097/01.hjr.0000096541.30533.82. PMID 14663300
- [Background] Nielsen EM, Hansen L, Echwald SM, Drivsholm T, Borch-Johnsen K, Ekstrom CT, Hansen T, Pedersen O. Evidence for an association between the Leu162Val polymorphism of the PPARalpha gene and decreased fasting serum triglyceride levels in glucose tolerant subjects. Pharmacogenetics. 2003 Jul;13(7):417-23. doi: 10.1097/01.fpc.0000054105.48725.5c. PMID 12835617
- [Background] Glumer C, Carstensen B, Sandbaek A, Lauritzen T, Jorgensen T, Borch-Johnsen K; inter99 study. A Danish diabetes risk score for targeted screening: the Inter99 study. Diabetes Care. 2004 Mar;27(3):727-33. doi: 10.2337/diacare.27.3.727. PMID 14988293
- [Background] Glumer C, Jorgensen T, Borch-Johnsen K. Targeted screening for undiagnosed diabetes reduces the number of diagnostic tests. Inter99(8). Diabet Med. 2004 Aug;21(8):874-80. doi: 10.1111/j.1464-5491.2004.01260.x. PMID 15270791
- [Background] Hansen SK, Gjesing AP, Rasmussen SK, Glumer C, Urhammer SA, Andersen G, Rose CS, Drivsholm T, Torekov SK, Jensen DP, Ekstrom CT, Borch-Johnsen K, Jorgensen T, McCarthy MI, Hansen T, Pedersen O. Large-scale studies of the HphI insulin gene variable-number-of-tandem-repeats polymorphism in relation to Type 2 diabetes mellitus and insulin release. Diabetologia. 2004 Jun;47(6):1079-87. doi: 10.1007/s00125-004-1418-3. Epub 2004 May 29. PMID 15170498
- [Background] Johansen A, Nielsen EM, Andersen G, Hamid YH, Jensen DP, Glumer C, Drivsholm T, Borch-Johnsen K, Jorgensen T, Hansen T, Pedersen O. Large-scale studies of the functional K variant of the butyrylcholinesterase gene in relation to Type 2 diabetes and insulin secretion. Diabetologia. 2004 Aug;47(8):1437-41. doi: 10.1007/s00125-004-1459-7. Epub 2004 Jul 17. PMID 15258737
- [Background] Andersen KL, Echwald SM, Larsen LH, Hamid YH, Glumer C, Jorgensen T, Borch-Johnsen K, Andersen T, Sorensen TI, Hansen T, Pedersen O. Variation of the McKusick-Kaufman gene and studies of relationships with common forms of obesity. J Clin Endocrinol Metab. 2005 Jan;90(1):225-30. doi: 10.1210/jc.2004-0465. Epub 2004 Oct 13. PMID 15483080
- [Background] Husemoen LL, Thomsen TF, Fenger M, Jorgensen T. Effect of lifestyle factors on plasma total homocysteine concentrations in relation to MTHFR(C677T) genotype. Inter99 (7). Eur J Clin Nutr. 2004 Aug;58(8):1142-50. doi: 10.1038/sj.ejcn.1601942. PMID 15054427
- [Background] Kessel L, Hougaard JL, Mortensen C, Jorgensen T, Lund-Andersen H, Larsen M. Visual acuity and refractive errors in a suburban Danish population: Inter99 Eye Study. Acta Ophthalmol Scand. 2004 Feb;82(1):19-24. doi: 10.1111/j.1395-3907.2004.0179.x. PMID 14738485
- [Background] Andersen G, Wegner L, Yanagisawa K, Rose CS, Lin J, Glumer C, Drivsholm T, Borch-Johnsen K, Jorgensen T, Hansen T, Spiegelman BM, Pedersen O. Evidence of an association between genetic variation of the coactivator PGC-1beta and obesity. J Med Genet. 2005 May;42(5):402-7. doi: 10.1136/jmg.2004.026278. PMID 15863669
- [Background] Andersen G, Wegner L, Jensen DP, Glumer C, Tarnow L, Drivsholm T, Poulsen P, Hansen SK, Nielsen EM, Ek J, Mouritzen P, Vaag A, Parving HH, Borch-Johnsen K, Jorgensen T, Hansen T, Pedersen O. PGC-1alpha Gly482Ser polymorphism associates with hypertension among Danish whites. Hypertension. 2005 Apr;45(4):565-70. doi: 10.1161/01.HYP.0000158946.53289.24. Epub 2005 Feb 28. PMID 15738346
- [Background] Hansen SK, Nielsen EM, Ek J, Andersen G, Glumer C, Carstensen B, Mouritzen P, Drivsholm T, Borch-Johnsen K, Jorgensen T, Hansen T, Pedersen O. Analysis of separate and combined effects of common variation in KCNJ11 and PPARG on risk of type 2 diabetes. J Clin Endocrinol Metab. 2005 Jun;90(6):3629-37. doi: 10.1210/jc.2004-1942. Epub 2005 Mar 29. PMID 15797964
- [Background] Rose CS, Andersen G, Hamid YH, Glumer C, Drivsholm T, Borch-Johnsen K, Jorgensen T, Pedersen O, Hansen T. Studies of relationships between the GLUT10 Ala206Thr polymorphism and impaired insulin secretion. Diabet Med. 2005 Jul;22(7):946-9. doi: 10.1111/j.1464-5491.2005.01547.x. PMID 15975113
- [Background] Ek J, Rose CS, Jensen DP, Glumer C, Borch-Johnsen K, Jorgensen T, Pedersen O, Hansen T. The functional Thr130Ile and Val255Met polymorphisms of the hepatocyte nuclear factor-4alpha (HNF4A): gene associations with type 2 diabetes or altered beta-cell function among Danes. J Clin Endocrinol Metab. 2005 May;90(5):3054-9. doi: 10.1210/jc.2004-2159. Epub 2005 Feb 22. PMID 15728204
- [Background] Faerch K, Lau C, Tetens I, Pedersen OB, Jorgensen T, Borch-Johnsen K, Glumer C. A statistical approach based on substitution of macronutrients provides additional information to models analyzing single dietary factors in relation to type 2 diabetes in danish adults: the Inter99 study. J Nutr. 2005 May;135(5):1177-82. doi: 10.1093/jn/135.5.1177. PMID 15867300
- [Background] Lau C, Faerch K, Glumer C, Tetens I, Pedersen O, Carstensen B, Jorgensen T, Borch-Johnsen K; Inter99 study. Dietary glycemic index, glycemic load, fiber, simple sugars, and insulin resistance: the Inter99 study. Diabetes Care. 2005 Jun;28(6):1397-403. doi: 10.2337/diacare.28.6.1397. PMID 15920058
- [Background] Glumer C, Borch-Johnsen K, Colagiuri S. Can a screening programme for diabetes be applied to another population? Diabet Med. 2005 Sep;22(9):1234-8. doi: 10.1111/j.1464-5491.2005.01641.x. PMID 16108854
- [Background] Hamid YH, Rose CS, Urhammer SA, Glumer C, Nolsoe R, Kristiansen OP, Mandrup-Poulsen T, Borch-Johnsen K, Jorgensen T, Hansen T, Pedersen O. Variations of the interleukin-6 promoter are associated with features of the metabolic syndrome in Caucasian Danes. Diabetologia. 2005 Feb;48(2):251-60. doi: 10.1007/s00125-004-1623-0. Epub 2005 Jan 11. PMID 15645209
- [Background] Hamid YH, Vissing H, Holst B, Urhammer SA, Pyke C, Hansen SK, Glumer C, Borch-Johnsen K, Jorgensen T, Schwartz TW, Pedersen O, Hansen T. Studies of relationships between variation of the human G protein-coupled receptor 40 Gene and Type 2 diabetes and insulin release. Diabet Med. 2005 Jan;22(1):74-80. doi: 10.1111/j.1464-5491.2005.01505.x. PMID 15606695
- [Background] Hamid YH, Urhammer SA, Glumer C, Borch-Johnsen K, Jorgensen T, Hansen T, Pedersen O. The common T60N polymorphism of the lymphotoxin-alpha gene is associated with type 2 diabetes and other phenotypes of the metabolic syndrome. Diabetologia. 2005 Mar;48(3):445-51. doi: 10.1007/s00125-004-1659-1. Epub 2005 Feb 24. PMID 15729581
- [Background] Hansen SK, Rose CS, Glumer C, Drivsholm T, Borch-Johnsen K, Jorgensen T, Pedersen O, Hansen T. Variation near the hepatocyte nuclear factor (HNF)-4alpha gene associates with type 2 diabetes in the Danish population. Diabetologia. 2005 Mar;48(3):452-8. doi: 10.1007/s00125-005-1671-0. Epub 2005 Feb 25. PMID 15735891
- [Background] Pisinger C, Vestbo J, Borch-Johnsen K, Thomsen T, Jorgensen T. Acceptance of the smoking cessation intervention in a large population-based study: the Inter99 study. Scand J Public Health. 2005;33(2):138-45. doi: 10.1080/14034940410028370. PMID 15823975
- [Background] Pisinger C, Vestbo J, Borch-Johnsen K, Jorgensen T. Smoking cessation intervention in a large randomised population-based study. The Inter99 study. Prev Med. 2005 Mar;40(3):285-92. doi: 10.1016/j.ypmed.2004.06.001. PMID 15533541
- [Background] Pisinger C, Vestbo J, Borch-Johnsen K, Jorgensen T. It is possible to help smokers in early motivational stages to quit. The Inter99 study. Prev Med. 2005 Mar;40(3):278-84. doi: 10.1016/j.ypmed.2004.06.011. PMID 15533540
- [Background] Pisinger C, Vestbo J, Borch-Johnsen K, Jorgensen T. Smoking reduction intervention in a large population-based study. The Inter99 study. Prev Med. 2005 Jan;40(1):112-8. doi: 10.1016/j.ypmed.2004.05.014. PMID 15530588
- [Background] Torekov SS, Larsen LH, Glumer C, Borch-Johnsen K, Jorgensen T, Holst JJ, Madsen OD, Hansen T, Pedersen O. Evidence of an association between the Arg72 allele of the peptide YY and increased risk of type 2 diabetes. Diabetes. 2005 Jul;54(7):2261-5. doi: 10.2337/diabetes.54.7.2261. PMID 15983231
- [Derived] Engelbrechtsen L, Mahendran Y, Jonsson A, Gjesing AP, Weeke PE, Jorgensen ME, Faerch K, Witte DR, Holst JJ, Jorgensen T, Grarup N, Pedersen O, Vestergaard H, Torekov S, Kanters JK, Hansen T. Common variants in the hERG (KCNH2) voltage-gated potassium channel are associated with altered fasting and glucose-stimulated plasma incretin and glucagon responses. BMC Genet. 2018 Mar 16;19(1):15. doi: 10.1186/s12863-018-0602-2. PMID 29548277
- [Derived] Svendstrup M, Appel EVR, Sandholt CH, Ahluwalia TS, Angquist LH, Thuesen BH, Jorgensen ME, Pedersen O, Grarup N, Hansen T, Sorensen TIA, Vestergaard H. Prospective Studies Exploring the Possible Impact of an ID3 Polymorphism on Changes in Obesity Measures. Obesity (Silver Spring). 2018 Apr;26(4):747-754. doi: 10.1002/oby.22109. Epub 2018 Feb 14. PMID 29442437
- [Derived] Hansen L, Netterstrom MK, Johansen NB, Ronn PF, Vistisen D, Husemoen LLN, Jorgensen ME, Rod NH, Faerch K. Metabolically Healthy Obesity and Ischemic Heart Disease: A 10-Year Follow-Up of the Inter99 Study. J Clin Endocrinol Metab. 2017 Jun 1;102(6):1934-1942. doi: 10.1210/jc.2016-3346. PMID 28323999
- [Derived] Ahluwalia TS, Troelsen JT, Balslev-Harder M, Bork-Jensen J, Thuesen BH, Cerqueira C, Linneberg A, Grarup N, Pedersen O, Hansen T, Dalgaard LT. Carriers of a VEGFA enhancer polymorphism selectively binding CHOP/DDIT3 are predisposed to increased circulating levels of thyroid-stimulating hormone. J Med Genet. 2017 Mar;54(3):166-175. doi: 10.1136/jmedgenet-2016-104084. Epub 2016 Sep 14. PMID 27627987
- [Derived] Lau CJ, Pisinger C, Husemoen LLN, Jacobsen RK, Linneberg A, Jorgensen T, Glumer C. Effect of general health screening and lifestyle counselling on incidence of diabetes in general population: Inter99 randomised trial. Prev Med. 2016 Oct;91:172-179. doi: 10.1016/j.ypmed.2016.08.016. Epub 2016 Aug 8. PMID 27514243
- [Derived] Bender AM, Jorgensen T, Pisinger C. Effects of general health checks differ under two different analyses perspectives-the Inter99 randomized study. J Clin Epidemiol. 2016 Mar;71:120-2. doi: 10.1016/j.jclinepi.2015.11.008. Epub 2015 Nov 18. No abstract available. PMID 26597976
- [Derived] Bender AM, Kawachi I, Jorgensen T, Pisinger C. Neighborhood social capital is associated with participation in health checks of a general population: a multilevel analysis of a population-based lifestyle intervention- the Inter99 study. BMC Public Health. 2015 Jul 22;15:694. doi: 10.1186/s12889-015-2042-5. PMID 26197982
- [Derived] Baumann S, Toft U, Aadahl M, Jorgensen T, Pisinger C. The long-term effect of screening and lifestyle counseling on changes in physical activity and diet: the Inter99 Study - a randomized controlled trial. Int J Behav Nutr Phys Act. 2015 Mar 6;12:33. doi: 10.1186/s12966-015-0195-3. PMID 25886540
- [Derived] Krarup NT, Borglykke A, Allin KH, Sandholt CH, Justesen JM, Andersson EA, Grarup N, Jorgensen T, Pedersen O, Hansen T. A genetic risk score of 45 coronary artery disease risk variants associates with increased risk of myocardial infarction in 6041 Danish individuals. Atherosclerosis. 2015 Jun;240(2):305-10. doi: 10.1016/j.atherosclerosis.2015.03.022. Epub 2015 Mar 16. PMID 25864160
- [Derived] Dashti HS, Follis JL, Smith CE, Tanaka T, Cade BE, Gottlieb DJ, Hruby A, Jacques PF, Lamon-Fava S, Richardson K, Saxena R, Scheer FA, Kovanen L, Bartz TM, Perala MM, Jonsson A, Frazier-Wood AC, Kalafati IP, Mikkila V, Partonen T, Lemaitre RN, Lahti J, Hernandez DG, Toft U, Johnson WC, Kanoni S, Raitakari OT, Perola M, Psaty BM, Ferrucci L, Grarup N, Highland HM, Rallidis L, Kahonen M, Havulinna AS, Siscovick DS, Raikkonen K, Jorgensen T, Rotter JI, Deloukas P, Viikari JS, Mozaffarian D, Linneberg A, Seppala I, Hansen T, Salomaa V, Gharib SA, Eriksson JG, Bandinelli S, Pedersen O, Rich SS, Dedoussis G, Lehtimaki T, Ordovas JM. Habitual sleep duration is associated with BMI and macronutrient intake and may be modified by CLOCK genetic variants. Am J Clin Nutr. 2015 Jan;101(1):135-43. doi: 10.3945/ajcn.114.095026. Epub 2014 Nov 26. PMID 25527757
- [Derived] Skaaby T, Nystrup Husemoen LL, Roswall N, Thuesen BH, Linneberg A. Atopy and development of cancer: a population-based prospective study. J Allergy Clin Immunol Pract. 2014 Nov-Dec;2(6):779-85. doi: 10.1016/j.jaip.2014.06.010. Epub 2014 Aug 28. PMID 25439371
- [Derived] Aadahl M, Linneberg A, Moller TC, Rosenorn S, Dunstan DW, Witte DR, Jorgensen T. Motivational counseling to reduce sitting time: a community-based randomized controlled trial in adults. Am J Prev Med. 2014 Nov;47(5):576-86. doi: 10.1016/j.amepre.2014.06.020. Epub 2014 Aug 8. PMID 25113139
- [Derived] Jorgensen T, Jacobsen RK, Toft U, Aadahl M, Glumer C, Pisinger C. Effect of screening and lifestyle counselling on incidence of ischaemic heart disease in general population: Inter99 randomised trial. BMJ. 2014 Jun 9;348:g3617. doi: 10.1136/bmj.g3617. PMID 24912589
- [Derived] Larsen SC, Angquist L, Ahluwalia TS, Skaaby T, Roswall N, Tjonneland A, Halkjaer J, Overvad K, Pedersen O, Hansen T, Linneberg A, Husemoen LL, Toft U, Heitmann BL, Sorensen TI. Dietary ascorbic acid and subsequent change in body weight and waist circumference: associations may depend on genetic predisposition to obesity--a prospective study of three independent cohorts. Nutr J. 2014 May 3;13:43. doi: 10.1186/1475-2891-13-43. PMID 24886192
- [Derived] Larsen SC, Angquist L, Ahluwalia TS, Skaaby T, Roswall N, Tjonneland A, Halkjaer J, Overvad K, Pedersen O, Hansen T, Linneberg A, Husemoen LL, Toft U, Heitmann BL, Sorensen TIa. Interaction between genetic predisposition to obesity and dietary calcium in relation to subsequent change in body weight and waist circumference. Am J Clin Nutr. 2014 Apr;99(4):957-65. doi: 10.3945/ajcn.113.076596. Epub 2014 Feb 5. PMID 24500147
- [Derived] Munch IC, Linneberg A, Larsen M. Precursors of age-related macular degeneration: associations with physical activity, obesity, and serum lipids in the inter99 eye study. Invest Ophthalmol Vis Sci. 2013 Jun 6;54(6):3932-40. doi: 10.1167/iovs.12-10785. PMID 23652489
- [Derived] Toft U, Jakobsen M, Aadahl M, Pisinger C, Jorgensen T. Does a population-based multi-factorial lifestyle intervention increase social inequality in dietary habits? The Inter99 study. Prev Med. 2012 Jan;54(1):88-93. doi: 10.1016/j.ypmed.2011.10.005. Epub 2011 Oct 15. PMID 22036837
- [Derived] Burgdorf KS, Gjesing AP, Grarup N, Justesen JM, Sandholt CH, Witte DR, Jorgensen T, Madsbad S, Hansen T, Pedersen O. Association studies of novel obesity-related gene variants with quantitative metabolic phenotypes in a population-based sample of 6,039 Danish individuals. Diabetologia. 2012 Jan;55(1):105-13. doi: 10.1007/s00125-011-2320-4. Epub 2011 Sep 28. PMID 21953277
- [Derived] Pilgaard K, Faerch K, Carstensen B, Poulsen P, Pisinger C, Pedersen O, Witte DR, Hansen T, Jorgensen T, Vaag A. Low birthweight and premature birth are both associated with type 2 diabetes in a random sample of middle-aged Danes. Diabetologia. 2010 Dec;53(12):2526-30. doi: 10.1007/s00125-010-1917-3. Epub 2010 Sep 22. PMID 20859612
- [Derived] Faerch K, Borch-Johnsen K, Vaag A, Jorgensen T, Witte DR. Sex differences in glucose levels: a consequence of physiology or methodological convenience? The Inter99 study. Diabetologia. 2010 May;53(5):858-65. doi: 10.1007/s00125-010-1673-4. Epub 2010 Feb 25. PMID 20182862
- [Derived] Munch IC, Ek J, Kessel L, Sander B, Almind GJ, Brondum-Nielsen K, Linneberg A, Larsen M. Small, hard macular drusen and peripheral drusen: associations with AMD genotypes in the Inter99 Eye Study. Invest Ophthalmol Vis Sci. 2010 May;51(5):2317-21. doi: 10.1167/iovs.09-4482. Epub 2009 Dec 10. PMID 20007824
- [Derived] Engberg S, Glumer C, Witte DR, Jorgensen T, Borch-Johnsen K. Differential relationship between physical activity and progression to diabetes by glucose tolerance status: the Inter99 Study. Diabetologia. 2010 Jan;53(1):70-8. doi: 10.1007/s00125-009-1587-1. Epub 2009 Nov 7. PMID 19898830
- [Derived] Engberg S, Vistisen D, Lau C, Glumer C, Jorgensen T, Pedersen O, Borch-Johnsen K. Progression to impaired glucose regulation and diabetes in the population-based Inter99 study. Diabetes Care. 2009 Apr;32(4):606-11. doi: 10.2337/dc08-1869. Epub 2008 Dec 29. PMID 19114617
- [Derived] Toft U, Kristoffersen L, Ladelund S, Ovesen L, Lau C, Pisinger C, Smith Lv, Borch-Johnsen K, Jorgensen T. The effect of adding group-based counselling to individual lifestyle counselling on changes in dietary intake. The Inter99 study--a randomized controlled trial. Int J Behav Nutr Phys Act. 2008 Nov 21;5:59. doi: 10.1186/1479-5868-5-59. PMID 19025583
- [Derived] Grarup N, Albrechtsen A, Ek J, Borch-Johnsen K, Jorgensen T, Schmitz O, Hansen T, Pedersen O. Variation in the peroxisome proliferator-activated receptor delta gene in relation to common metabolic traits in 7,495 middle-aged white people. Diabetologia. 2007 Jun;50(6):1201-8. doi: 10.1007/s00125-007-0668-2. Epub 2007 Apr 13. PMID 17431579
- See also: Study description and results. All publications available. Also in English. — http://www.Inter99.dk